CLINICAL TRIAL: NCT03907267
Title: Taurine for Early Left Ventricular Recovery in Peripartum Cardiomyopathy
Brief Title: Taurine in Peripartum Cardiomyopathy
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Mohamed S Sweed, MD, Principal Investigator, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AS1755
Record Dates: First submitted 2019-04-05; First posted 2019-04-08 (Actual); Last update posted 2020-01-28 (Actual); Status verified 2020-01

CONDITIONS: Peripartum Cardiomyopathy
MeSH Terms: conditions — Peripartum Cardiomyopathy | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Taurine (Experimental)
  Interventions: Drug: Taurine Solution
- Saline (Placebo Comparator)
  Interventions: Dietary Supplement: Normal Saline

INTERVENTIONS:
Drug: Taurine Solution — Taurine Solution
  Arms: Taurine
Dietary Supplement: Normal Saline — Normal Saline
  Arms: Saline

SUMMARY:
Taurine as an adjunct for early left ventricular recovery in peripartum cardiomyopathy

ELIGIBILITY:
Inclusion Criteria:

* Peripartum Cardiomyopathy

Exclusion Criteria:

* Other identifiable cause for heart failure
* low LVEF ≤ 25%
* sepsis
* autoimmune disease
* severe chronic disease
* malignancy

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2020-01-01 (Actual)

PRIMARY OUTCOMES:
improvement of the left ventricular ejection fraction >10 % | 1 week
  improvement of the left ventricular ejection fraction >10 %

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University Maternity Hospital, Cairo, Egypt